CLINICAL TRIAL: NCT06277947
Title: Administration of Hyperthermic Intraperitoneal Chemotherapy in the General Ward: a Multicenter, Prospective, Feasibility Study (GARD-HIPEC Study)
Brief Title: Administration of Hyperthermic Intraperitoneal Chemotherapy in the General Ward
Acronym: GARD-HIPEC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Shenshan Medical Center, Memorial Hospital of Sun Yat-sen University (Unknown)
Responsible Party: Principal Investigator, Jing Li, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-096-01
Record Dates: First submitted 2024-02-03; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer; Hyperthermic Intraperitoneal Chemotherapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Intervention Model Description: Patients would receive C-HIPEC in the general ward after interval debulking surgery in 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-HIPEC arm (Experimental): Infuse paclitaxel (75mg/m^2) and cisplatin (75mg/m^2) at 43℃ through the two drainage tubes placed in the upper abdomen, using the two drainage tubes placed in the lower abdomen as the effluent tubes, with an infusion time of 90 minutes and an infusion rate of 500-600 mL/min. The first HIPEC with paclitaxel should be performed within 24 hours after cytoreductive surgery. The second HIPEC with cisplatin should be performed 24 hours after the completion of the first HIPEC. Intravenous sedatives such as diazoxide, or propofol at 2-6 ml/h should be administered during HIPEC treatment with continuous intravenous infusion by a pump，or intramuscular injection of 50 mg of pethidine.
  Interventions: Procedure: China Hyperthermic Intraperitoneal Chemotherapy(C-HIPEC)

INTERVENTIONS:
Procedure: China Hyperthermic Intraperitoneal Chemotherapy(C-HIPEC) — The C-HIPEC would be performed at bedside in the general ward within 24 hours after surgery. The HIPEC treatment instruments are BR-TRG-II system, which can control the temperature stably to 43℃±0.1℃.

SUMMARY:
Ovarian cancer is the most lethal gynecologic malignancy. The majority of patients get diagnosed with advanced disease with peritoneal dissemination.It has been demonstrated that the addition of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) to interval debulking surgery can improve the prognosis. The National Comprehensive Cancer Network (NCCN) treatment guideline has recommended HIPEC as a first-line treatment for patients with advanced ovarian cancer. However, the guideline recommended the "Dutch model" of HIPEC, which is limited for routinely being performed in China. So we propose a HIPEC treatment modality, the bedside closed HIPEC in the general ward (C-HIPEC), which is suitable for the clinical characteristics of China. The aim of this study was to evaluate the safety of this model as a way to lay the foundation for subsequent efficacy evaluation and clinical promotion.

DETAILED DESCRIPTION:
The Dutch Model is limited for the following reasons: 1) The HIPEC treatment requires to be done in the operating room, which means the operation time would be lengthened. 2) High rate of exposure to chemotherapeutic drugs among healthcare workers. 3) It has significant safety concerns because it does not take into account racial differences in drug toxicity. This study is an investigator-initiated prospective multicenter feasibility study with a non-inferiority design, so as to provide evidence-based medical evidence for the use of the C-HIPEC model as an alternative to the "Dutch model" in clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:（The following conditions must be met at the same time）

1. Pathologically confirmed primary epithelial ovarian, fallopian tube, and primary peritoneal cancers in FIGO stages III-IV.
2. Previous neoadjuvant chemotherapy with platinum + vincristine and ≤ 4 courses of neoadjuvant chemotherapy.
3. The residual tumor diameter is ≤1 cm after interval debulking surgery, and the reason for receiving IDS is that the patient cannot tolerate PDS due to the poor condition or the PDS cannot achieve optimal cytoreduction due to high tumor burden.
4. Age from 18 to 70 years.
5. Bone marrow reserve was well functioning. Leukocytosis ≥ 3.0×10^9/L, neutrophilic granulocyte ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, and hemoglobin ≥ 80 g/L.
6. Organs work well. AST ≤ 2.5 × ULN, ALT ≤ 2.5 × upper limit of normal(ULN), total serum bilirubin ≤ 1.5 × ULN, and creatinine ≤ 1.5 × ULN.
7. ECOG score 0-1.
8. Patients voluntarily sign an informed consent form

Exclusion Criteria: (None of which was eligible)

1. Patients diagnosed with other malignant tumors within 5 years (excluding skin and thyroid cancers).
2. Patient is allergic to erythroxylanes.
3. Patients treated with anticancer drugs in other clinical trials.
4. High risk of anastomotic fistula or intestinal obstruction assessed during interval debulking surgery.
5. Any situation of disease instability or potentially impact safety and adherence of patient.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events of grade 3-5 | up to 3 weeks after C-HIPEC.
  The adverse events would be graded according to Common Terminology Criteria for Adverse Events (CTCAE 5.0). The types and incidence of AEs will be recorded to evaluate the safety of C-HIPEC.

SECONDARY OUTCOMES:
Time to progress (TTP) | from the end of IV chemotherapy to 1 year after C-HIPEC or relapse
  Disease progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1, or on the basis of an increase from baseline in the CA-125 level, whichever one of these two criteria was met first. The CA-125 will be tested before each chemotherapy session, and the radiographic examination will be done every 3 months since the end of IV chemotherapy.
The Time to the First Subsequent Therapy，TTFST | C-HIPEC to the first subsequent IV chemotherapy
  The Time to the First Subsequent Therapy
Quality of life, QLQ-C30 | 1) within 2 weeks before C-HIPEC; 2) 1 week after C-HIPEC; 3) before each cycle of IV chemotherapy (each cycle is 28 days)
  Quality of life is assessed by health-related quality-of-life questionnaires-the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledermann JA, Raja FA, Fotopoulou C, Gonzalez-Martin A, Colombo N, Sessa C; ESMO Guidelines Working Group. Newly diagnosed and relapsed epithelial ovarian carcinoma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi24-32. doi: 10.1093/annonc/mdt333. No abstract available. PMID 24078660
- [Background] Sin EI, Chia CS, Tan GHC, Soo KC, Teo MC. Acute kidney injury in ovarian cancer patients undergoing cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy. Int J Hyperthermia. 2017 Sep;33(6):690-695. doi: 10.1080/02656736.2017.1293304. Epub 2017 Mar 5. PMID 28540777
- [Background] Chambers LM, Costales AB, Crean-Tate K, Kuznicki M, Morton M, Horowitz M, Jagielo T, Rose PG, Michener C, Vargas R, Debernardo R. A guide to establishing a hyperthermic intraperitoneal chemotherapy program in gynecologic oncology. Gynecol Oncol. 2020 Sep;158(3):794-802. doi: 10.1016/j.ygyno.2020.06.487. Epub 2020 Jul 2. PMID 32624234
- [Background] Lemoine L, Sugarbaker P, Van der Speeten K. Drugs, doses, and durations of intraperitoneal chemotherapy: standardising HIPEC and EPIC for colorectal, appendiceal, gastric, ovarian peritoneal surface malignancies and peritoneal mesothelioma. Int J Hyperthermia. 2017 Aug;33(5):582-592. doi: 10.1080/02656736.2017.1291999. PMID 28540826
- [Background] Wu MF, Cheng XY, Wang DY, Lai YT, Li H, Ye YF, Peng YP, Chen Q, Zhang BZ, Lin ZQ, Li J. Determining the maximum tolerated dose of paclitaxel combined with fixed dose of cisplatin for hyperthermic intraperitoneal chemotherapy in ovarian cancer: A multicenter phase I trial. Gynecol Oncol. 2024 Feb;181:125-132. doi: 10.1016/j.ygyno.2023.12.019. Epub 2023 Dec 30. PMID 38159362
- [Result] Arjona-Sanchez A, Espinosa-Redondo E, Gutierrez-Calvo A, Segura-Sampedro JJ, Perez-Viejo E, Concepcion-Martin V, Sanchez-Garcia S, Garcia-Fadrique A, Prieto-Nieto I, Barrios-Sanchez P, Torres-Melero J, Ramirez Faraco M, Prada-Villaverde A, Carrasco-Campos J, Artiles-Armas M, Villarejo-Campos P, Ortega-Perez G, Boldo-Roda E, Sanchez-Hidalgo JM, Casado-Adam A, Rodriguez-Ortiz L, Aranda E, Cano-Osuna MT, Diaz-Lopez C, Romero-Ruiz A, Briceno-Delgado J, Rufian-Pena S; Grupo Espanol de Carcinomatosis Peritoneal. Efficacy and Safety of Intraoperative Hyperthermic Intraperitoneal Chemotherapy for Locally Advanced Colon Cancer: A Phase 3 Randomized Clinical Trial. JAMA Surg. 2023 Jul 1;158(7):683-691. doi: 10.1001/jamasurg.2023.0662. PMID 37099280
- [Result] Lee JY, Lee YJ, Son JH, Kim S, Choi MC, Suh DH, Song JY, Hong DG, Kim MK, Kim JH, Chang SJ. Hyperthermic Intraperitoneal Chemotherapy After Interval Cytoreductive Surgery for Patients With Advanced-Stage Ovarian Cancer Who Had Received Neoadjuvant Chemotherapy. JAMA Surg. 2023 Nov 1;158(11):1133-1140. doi: 10.1001/jamasurg.2023.3944. PMID 37672264
- [Result] Lim MC, Chang SJ, Park B, Yoo HJ, Yoo CW, Nam BH, Park SY; HIPEC for Ovarian Cancer Collaborators. Survival After Hyperthermic Intraperitoneal Chemotherapy and Primary or Interval Cytoreductive Surgery in Ovarian Cancer: A Randomized Clinical Trial. JAMA Surg. 2022 May 1;157(5):374-383. doi: 10.1001/jamasurg.2022.0143. PMID 35262624
- [Result] Aronson SL, Lopez-Yurda M, Koole SN, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van Gent MDJM, Arts HJG, van Ham MAPC, van Dam PA, Vuylsteke P, Aalbers AGJ, Verwaal VJ, Van de Vijver KK, Aaronson NK, Sonke GS, van Driel WJ. Cytoreductive surgery with or without hyperthermic intraperitoneal chemotherapy in patients with advanced ovarian cancer (OVHIPEC-1): final survival analysis of a randomised, controlled, phase 3 trial. Lancet Oncol. 2023 Oct;24(10):1109-1118. doi: 10.1016/S1470-2045(23)00396-0. Epub 2023 Sep 11. PMID 37708912
- [Result] Chan CY, Li H, Wu MF, Liu CH, Lu HW, Lin ZQ, Li J. A Dose-Finding Trial for Hyperthermic Intraperitoneal Cisplatin in Gynecological Cancer Patients Receiving Hyperthermic Intraperitoneal Chemotherapy. Front Oncol. 2021 Mar 11;11:616264. doi: 10.3389/fonc.2021.616264. eCollection 2021. PMID 33777754
- [Result] You ZY, Wu MF, Li H, Ye YF, Wang LJ, Lin ZQ, Li J. A phase I dose-finding trial of hyperthermic intraperitoneal docetaxel combined with cisplatin in patients with advanced-stage ovarian cancer. J Gynecol Oncol. 2024 Jan;35(1):e1. doi: 10.3802/jgo.2024.35.e1. Epub 2023 Jul 5. PMID 37477105